CLINICAL TRIAL: NCT05133544
Title: Endocuff With or Without Artificial Intelligence-assisted Colonoscopy in Detection of Colorectal Adenoma: a Randomized Colonoscopy Trial
Brief Title: Endocuff With or Without AI-assisted Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Lui Ka-Luen, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: UW 20-647
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Colonic Adenoma; Colonic Polyp; Colonic Cancer
Keywords: Artificial intelligence; Colonoscopy; Endocuff; Detection; Computer-aided
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Endocuff- AI assisted colonoscopy (Active Comparator): Endocuff (Olympus, Hong Kong) and AI assisted colonoscopy will be used
  Interventions: Device: Endocuff with AI
- AI-assisted colonoscopy (Active Comparator): AI assisted colonoscopy will be used
  Interventions: Device: AI alone
- Conventional colonoscopy (No Intervention): Conventional colonoscopy will be used without AI or Endocuff.

INTERVENTIONS:
Device: Endocuff with AI — Use of endocuff with computer assisted polyp detection
  Arms: Endocuff- AI assisted colonoscopy
Device: AI alone — Use of computer assisted polyp detection
  Arms: AI-assisted colonoscopy

SUMMARY:
Colonoscopy is considered the gold standard for diagnosis of colonic polyps. However, it was reported that colonoscopy could still miss colonic polyps. Many attempts have been made to improve the detection rate of colonoscopy. Artificial intelligence (AI) is a promising new technique to improve detection rate of colonic adenoma. However, it remains uncertain whether whether the combined use of Endocuff and AI assisted examination could help to further improve the adenoma detection rate. This is a prospective randomized trial comparing the use of endocuff with AI, AI alone or conventional colonoscopy examination on adenoma detection rate.

DETAILED DESCRIPTION:
TThis is a prospective randomized tandem colonoscopy trial comparing three different modes of colonoscopy techniques. The first group will use Endocuff (Olympus, Hong Kong) and AI assisted colonoscopy. The second group will use AI assisted colonoscopy alone and the third group will use standard high-definition white light colonoscopy.

Eligible patients will be randomly allocated in a 1:1:1 ratio to three groups. Patients will be stratified according to indications of colonoscopy (symptomatic vs screening/surveillance).

All examination will be performed with high-definition endoscopes (EVIS-EXERA 290 video system, Olympus Optical, Tokyo, Japan) under white light by experienced endoscopists. All endoscopists should have received training on the interpretation of real-time AI detection system as well as the Endocuff before performing study colonoscopy.

In all colonoscopy examination, colonoscope will be first advanced to the cecum as confirmed by identification of the appendiceal orifice and ileocecal valve or by intubation of the ileum. After cecal intubation is performed, the colonoscopy is first withdrawn according to the group assigned. For group 1, the first withdrawal would be done with Endocuff and AI assistance. For group 2, the first withdrawal would be done under AI assistance only. For group 3, the first withdrawal would be done under standard high definition colonoscopy only.

All detected polyps will be removed during the withdrawal only. The size (measured with biopsy forceps), location and morphology of each polyp will be recorded by an independent observer. The withdrawal time (minus the polypectomy site) will be measured by a stopwatch and with a minimum of 6 minutes. The bowel preparation quality will be graded according to the Boston Bowel Preparation Scale

ELIGIBILITY:
Inclusion Criteria:

* All adult patients, aged 40 or above, undergoing outpatient colonoscopy in the Queen Mary Hospital, Tung Wah Hospital and Tuen Mun Hospital in Hong Kong will be recruited.

Exclusion Criteria:

* Patients will be excluded if they have history of inflammatory bowel disease, colorectal cancer, previous bowel resection, Peutz-Jeghers syndrome, familial adenomatous polyposis or other polyposis syndromes, bleeding tendency or severe comorbid illnesses for which polypectomy is considered unsafe. Moreover, after randomization, if the cecum could not be intubated for various reasons or Boston Bowel Preparation Scale (BBPS) score is <2, these patients will be excluded

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 656 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | One month after colonoscopy
  The proportion of patients with at least one adenomas

SECONDARY OUTCOMES:
Polyp detection rate | One month after colonoscopy
  the proportion of patients with at least one polyp
Sessile serrated adenomas detection rate | One month after colonoscopy
  The proportion of patients with at least one sessile serrated adenomas
Sessile serrated polyps detection rate | One month after colonoscopy
  The proportion of patients with at least one sessile serrated polyps
Advanced adenoma detection rates | One month after colonoscopy
  The proportion of patients with at least one advanced adenomas
Mean number of polyp per patient | One month after colonoscopy
  The mean number of polyp per patient
Mean number of adenoma per patient | One month after colonoscopy
  The mean number of adenoma per patient
Total number of polyp or adenoma per patient. | One month after colonoscopy
  The total number of polyp or adenoma per patient.

CONTACTS AND LOCATIONS:
Overall Officials: Wai Keung Leung, MD, Study Director — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lui TK, Lam CP, To EW, Ko MK, Tsui VWM, Liu KS, Hui CK, Cheung MK, Mak LL, Hui RW, Wong SY, Seto WK, Leung WK. Endocuff With or Without Artificial Intelligence-Assisted Colonoscopy in Detection of Colorectal Adenoma: A Randomized Colonoscopy Trial. Am J Gastroenterol. 2024 Jul 1;119(7):1318-1325. doi: 10.14309/ajg.0000000000002684. Epub 2024 Feb 2. PMID 38305278